CLINICAL TRIAL: NCT04016714
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active-comparator-controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 3-dose Regimen of V114 in Healthy Infants (PNEU-PED-EU-2)
Brief Title: Safety, Tolerability, and Immunogenicity of a 3-dose Regimen of V114 in Healthy Infants (PNEU-PED-EU-2/V114-026)
Acronym: PNEU-PED-EU-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V114-026; V114-026 (Other: Merck Protocol Number); 2018-003788-70 (EudraCT Number)
Record Dates: First submitted 2019-07-10; First posted 2019-07-11 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; Vaxelis; Measles-Mumps-Rubella Vaccine; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 at Visit 1, 2, and 4 (approximately 3, 5, and 12 months of age). As part of the study design, participants will also receive other pediatric vaccines, including Vaxelis™ (0.5 mL single dose at Visits 1, 2, and 4); M-M-R™II (0.5 mL single dose at Visit 4); and VARIVAX™ (0.5 mL single dose at Visit 4, except participants in Norway and Denmark, who will receive a second dose of VARIVAX™ at Visit 5, according to local vaccination requirements).
  Interventions: Drug: V114; Drug: Vaxelis™; Drug: M-M-R®II; Drug: VARIVAX™
- Prevenar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevenar 13™ at Visit 1, 2, and 4 (approximately 3, 5, and 12 months of age). As part of the study design, participants will also receive other pediatric vaccines, including Vaxelis™ (0.5 mL single dose at Visits 1, 2, and 4); M-M-R™II (0.5 mL single dose at Visit 4); and VARIVAX™ (0.5 mL single dose at Visit 4, except participants in Norway and Denmark, who will receive a second dose of VARIVAX™ at Visit 5, according to local vaccination requirements).
  Interventions: Drug: Prevenar 13™; Drug: Vaxelis™; Drug: M-M-R®II; Drug: VARIVAX™

INTERVENTIONS:
Drug: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F, serotype 6B and aluminum phosphate adjuvant in each 0.5 mL dose.
  Other Names: VAXNEUVANCE™; Pneumococcal 15-Valent Conjugate Vaccine
  Arms: V114
Drug: Prevenar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F, serotype 6B in each 0.5. mL dose.
  Other Names: Prevnar 13™
  Arms: Prevenar 13™
Drug: Vaxelis™ — Intramuscular 0.5 mL single dose
Drug: M-M-R®II — Subcutaneous 0.5 mL single dose
  Other Names: Measles, Mumps, and Rubella Virus Vaccine Live
Drug: VARIVAX™ — Subcutaneous 0.5 mL single dose
  Other Names: Varicella Vaccine Live

SUMMARY:
The purpose of this clinical study is to evaluate the safety and immunogenicity of a 3-dose schedule (2-dose primary series followed by a toddler dose) of pneumococcal conjugate vaccine (PCV) as one of the currently recommended schedules by the World Health Organization (WHO) Strategic Advisory Group of Experts (SAGE) on Immunizations and practiced in many countries.

The primary hypotheses are that V114 is non-inferior to Prevenar 13™ for the 13 shared serotypes based on response rates and on anti-pneumococcal polysaccharide (PnPs) serotype-specific Immunoglobulin G (IgG) geometric mean concentrations (GMCs) at 30 days following Dose 3; that V114 is superior to Prevenar 13™ for the 2 serotypes unique to V114 based on the response rates and on anti-PnPs serotype-specific IgG GMCs at 30 days following Dose 3; and that Vaxelis™ administered concomitantly with V114 is non-inferior to Vaxelis™ administered concomitantly with Prevenar 13™ at 30 days following Dose 3 for each antigen included in Vaxelis™.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female, approximately 3 months of age, from 70 days to 111 days inclusive, at the time of signing the informed consent.
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria:

* Was born prior to 37 weeks of gestation.
* Has a history of invasive pneumococcal disease (IPD) or known history of other culture positive pneumococcal disease.
* Has a known hypersensitivity to any component of the pneumococcal conjugate vaccine (PCV), any component of the licensed pediatric vaccines to be administered concomitantly in the study, or any diphtheria toxoid containing vaccine.
* Has any contraindication to the concomitant study vaccines being administered in the study.
* Has a known or suspected impairment of immunological function.
* Has a history of congenital or acquired immunodeficiency.
* Has, or his/her mother has, a documented human immunodeficiency virus (HIV) infection.
* Has, or his/her mother has, a documented hepatitis B surface antigen - positive test.
* Has known or history of functional or anatomic asplenia.
* Has failure to thrive based on the clinical judgement of the investigator.
* Has a bleeding disorder contraindicating intramuscular vaccination.
* Has a history of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Behcet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, type 1 diabetes mellitus, or other autoimmune disorders).
* Has a known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders.
* Has received a dose of any pneumococcal vaccine prior to study entry.
* Has received >1 dose of monovalent hepatitis B vaccine or hepatitis B-based combination vaccine prior to study entry.
* Has received a dose of any acellular pertussis- or whole cell pertussis-based combination vaccines, Haemophilus influenza type b conjugate vaccine, poliovirus vaccine, or any other combination thereof, prior to study entry.
* Has received a blood transfusion or blood products, including immunoglobulins.
* Has participated in another clinical study of an investigational product before the beginning or anytime during the duration of the current clinical study. Participants enrolled in observational studies may be included; these will be reviewed on a case by-case basis for approval by the Sponsor.
* Has any other reason that, in the opinion of the investigator, may interfere with the evaluation required by the study. Reasons may include, but are not limited to, being unable to keep appointments or planning to relocate during the study.
* Is or has an immediate family member (e.g., parent/legal guardian or sibling) who is investigational site or Sponsor staff directly involved with this study.

Ages: 70 Days to 111 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1191 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (24):
- Denmark (6):
  - Hvidovre Hospital ( Site 0003), Hvidovre, Capital Region
  - Aarhus Universitetshosp. Skejby ( Site 0002), Aarhus, Central Jutland
  - Regionshospitalet Herning Hospitalsenheden Vest ( Site 0006), Herning, Central Jutland
  - Aalborg Universitetshospital ( Site 0005), Aalborg, North Denmark
  - Sygehus Vendsyssel Hjoerring ( Site 0004), Hjørring, North Denmark
  - Odense Universitetshospital ( Site 0001), Odense C, Region Syddanmark
- Finland (10):
  - Kokkolan rokotetutkimusklinikka ( Site 0029), Kokkola, Keski-Pohjanmaa
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 0030), Oulu, North Ostrobothnia
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 0021), Tampere, Pirkanmaa
  - Porin rokotetutkimusklinikka ( Site 0027), Pori, Satakunta
  - Seinajoki Vaccine Research Center ( Site 0028), Seinäjoki, South Ostrobothnia
  - Turun rokotetutkimuskeskus ( Site 0026), Turku, Southwest Finland
  - Tampereen yliopisto Espoon rokotetutkimusklinikka ( Site 0024), Espoo, Uusimaa
  - Tampereen yliopisto Etela-Helsingin Rokotetutkimusklinikka ( Site 0022), Helsinki, Uusimaa
  - Tampereen yliopisto Ita-Helsingin rokotetutkimusklinikka ( Site 0023), Helsinki, Uusimaa
  - Jarvenpaan rokotetutkimuskeskus ( Site 0025), Jarvenpaa, Uusimaa
- Italy (4):
  - Policlinico Universitario Agostino Gemelli ( Site 0048), Rome, Roma
  - A.O. Policlinico Consorziale di Bari ( Site 0044), Bari
  - A.O.U. Riuniti Di Foggia - Igiene Universitaria ( Site 0046), Foggia
  - IRCCS Ospedale Policlinico San Martino ( Site 0042), Genova
- Norway (3):
  - Stavanger universitetssykehus ( Site 0062), Stavanger, Rogaland
  - Sykehuset i Vestfold ( Site 0063), Tønsberg, Vestfold
  - Oslo Universitetssykehus HF Ulleval Sykehus ( Site 0061), Oslo
- Norrlands Universitetssjukhus ( Site 0100), Umeå, Vasterbottens Lan [se-24], Sweden

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Benfield T, Ramet M, Valentini P, Seppa I, Dagan R, Richmond P, Mercer S, Churchill C, Lupinacci R, McFetridge R, Park J, Wittke F, Banniettis N, Musey L, Bickham K, Kaminski J. Safety, tolerability, and immunogenicity of V114 pneumococcal vaccine compared with PCV13 in a 2+1 regimen in healthy infants: A phase III study (PNEU-PED-EU-2). Vaccine. 2023 Apr 6;41(15):2456-2465. doi: 10.1016/j.vaccine.2023.02.041. Epub 2023 Feb 24. PMID 36841723

RESULTS

PARTICIPANT FLOW:
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 at Visit 1, 2, and 4 (approximately 3, 5, and 12 months of age). As part of the study design, participants also received other pediatric vaccines, including Vaxelis™ (0.5 mL single dose at Visits 1, 2, and 4); M-M-R™II (0.5 mL single dose at Visit 4); and VARIVAX™ (0.5 mL single dose at Visit 4, except participants in Norway and Denmark, who received a second dose of VARIVAX™ at Visit 5, according to local vaccination requirements).
- Prevenar 13™: Participants received a single 0.5 mL IM injection of Prevenar 13™ at Visit 1, 2, and 4 (approximately 3, 5, and 12 months of age). As part of the study design, participants also received other pediatric vaccines, including Vaxelis™ (0.5 mL single dose at Visits 1, 2, and 4); M-M-R™II (0.5 mL single dose at Visit 4); and VARIVAX™ (0.5 mL single dose at Visit 4, except participants in Norway and Denmark, who received a second dose of VARIVAX™ at Visit 5, according to local vaccination requirements).
Period: Overall Study
Arm/Group | V114 | Prevenar 13™
Started | 595 | 596
Vaccination 1 (V114 or Prevenar 13™) | 595 | 596
Vaccination 2 (V114 or Prevenar 13™) | 585 | 588
Vaccination 3 (V114 or Prevenar 13™) | 573 | 581
Completed | 572 | 580
Not Completed | 23 | 16
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Parent/Guardian | 16 | 12

BASELINE CHARACTERISTICS:
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 at Visit 1, 2 and 4 (approximately 3, 5, and 12 months of age). As part of the study design, participants also received other pediatric vaccines, including Vaxelis™ (0.5 mL single dose at Visits 1, 2, and 4); M-M-R™II (0.5 mL single dose at Visit 4); and VARIVAX™ (0.5 mL single dose at Visit 4, except participants in Norway and Denmark, who received a second dose of VARIVAX™ at Visit 5, according to local vaccination requirements).
- Prevenar 13™: Participants received a single 0.5 mL IM injection of Prevenar 13™ at Visit 1, 2 and 4 (approximately 3, 5, and 12 months of age). As part of the study design, participants also received other pediatric vaccines, including Vaxelis™ (0.5 mL single dose at Visits 1, 2, and 4); M-M-R™II (0.5 mL single dose at Visit 4); and VARIVAX™ (0.5 mL single dose at Visit 4, except participants in Norway and Denmark, who received a second dose of VARIVAX™ at Visit 5, according to local vaccination requirements).
- Total: Total of all reporting groups
Arm/Group | V114 | Prevenar 13™ | Total
Number analyzed (Participants) | 595 | 596 | 1191
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 12.4 (1.4) | 12.5 (1.4) | 12.4 (1.4)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 595 | 596 | 1191
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 289 | 561
  Male | 323 | 307 | 630
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 579 | 579 | 1158
  More than one race | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 22 | 48
  Not Hispanic or Latino | 564 | 570 | 1134
  Not Reported | 3 | 3 | 6
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs included injection-site erythema (redness), injection-site induration (hard lump), injection-site pain (tenderness), and injection-site swelling.
Time Frame: Day 1 to Day 14 after each vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 595 | 594
Percentage of participants
  Injection-site erythema | 60.0 | 65.5
  Injection-site induration | 57.0 | 59.1
  Injection-site pain | 63.0 | 59.6
  Injection-site swelling | 46.4 | 44.1
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Injection-site erythema; Test type: Other; p = 0.050, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = -5.5, 95% CI 2-sided [-11.0 to 0.0]
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Injection-site induration; Test type: Other; p = 0.460, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = -2.1, 95% CI 2-sided [-7.7 to 3.5]
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Injection-site pain; Test type: Other; p = 0.225, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = 3.4, 95% CI 2-sided [-2.1 to 8.9]
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Injection-site swelling; Test type: Other; p = 0.430, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = 2.3, 95% CI 2-sided [-3.4 to 7.9]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs included decreased appetite, irritability, somnolence (drowsiness), and urticaria (hives or welts).
Time Frame: Day 1 to Day 14 after each vaccination
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 595 | 594
Percentage of participants
  Decreased appetite | 54.8 | 58.2
  Irritability | 96.3 | 94.1
  Somnolence | 77.3 | 77.9
  Urticaria | 16.8 | 21.4
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Decreased appetite; Test type: Other; p = 0.229, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = -3.5, 95% CI 2-sided [-9.1 to 2.2]
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Irritability; Test type: Other; p = 0.077, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = 2.2, 95% CI 2-sided [-0.2 to 4.7]
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Somnolence; Test type: Other; p = 0.793, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = -0.6, 95% CI 2-sided [-5.4 to 4.1]
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Urticaria; Test type: Other; p = 0.045, Miettinen & Nurminen method; Difference in percentage vs Prevenar 13™ = -4.6, 95% CI 2-sided [-9.1 to -0.1]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event
Description: A serious adverse event (SAE) is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. SAEs that were reported by the investigator to be at least possibly related to the study vaccination were summarized.
Time Frame: Up to approximately 6 months after Dose 3 (up to approximately 16 months)
Population: All randomized participants who received at least 1 dose of study vaccination
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 595 | 594
Percentage of participants | 0.3 | 0.3
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Vaccine-related SAEs; Test type: Other; Difference in percentage vs Prevenar 13™ = -0.0, 95% CI 2-sided [-0.9 to 0.9]

4. Primary Outcome: Percentage of Participants Meeting Serotype-specific Immunoglobulin G (IgG) Threshold Value of ≥0.35 μg/mL 30 Days After Dose 3
Description: The geometric mean concentration (GMC) of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevenar 13™ and 2 serotypes (22F and 33F) unique to V114 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay. Immunoglobulin G for the 15 serotypes contained in V114 vaccine was determined using a pneumococcal electrochemiluminescence (PnECL) assay.
Time Frame: 30 days after Dose 3
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and who had sufficient data to perform the analysis for each serotype
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 500 | 525
Percentage of participants
  Serotype 1 | 96.8 | 99.0
  Serotype 3 | 92.8 | 82.3
  Serotype 4: number analyzed (Participants) | 500 | 523
  Serotype 4 | 96.6 | 98.5
  Serotype 5: number analyzed (Participants) | 500 | 524
  Serotype 5 | 99.4 | 99.6
  Serotype 6A: number analyzed (Participants) | 500 | 523
  Serotype 6A | 99.2 | 99.4
  Serotype 6B: number analyzed (Participants) | 500 | 523
  Serotype 6B | 99.2 | 99.0
  Serotype 7F | 100.0 | 99.6
  Serotype 9V: number analyzed (Participants) | 499 | 525
  Serotype 9V | 99.8 | 99.6
  Serotype 14: number analyzed (Participants) | 500 | 523
  Serotype 14 | 99.2 | 99.6
  Serotype 18C | 99.8 | 99.4
  Serotype 19A: number analyzed (Participants) | 500 | 523
  Serotype 19A | 99.6 | 99.8
  Serotype 19F: number analyzed (Participants) | 500 | 524
  Serotype 19F | 99.8 | 99.6
  Serotype 23F: number analyzed (Participants) | 497 | 521
  Serotype 23F | 97.8 | 96.9
  Serotype 22F: number analyzed (Participants) | 500 | 520
  Serotype 22F | 99.4 | 5.4
  Serotype 33F: number analyzed (Participants) | 500 | 510
  Serotype 33F | 99.2 | 2.0
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Serotype 1; Test type: Non-Inferiority — For the 13 shared serotypes, a conclusion of non-inferiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% confidence interval (CI) for the difference in percentages (V114 - Prevenar 13™) being >-10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen method; Percentage point difference = -2.2, 95% CI 2-sided [-4.3 to -0.6]
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Serotype 3; Test type: Non-Inferiority — For the 13 shared serotypes, a conclusion of non-inferiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevenar 13™) being >-10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen method; Percentage point difference = 10.5, 95% CI 2-sided [6.6 to 14.6]
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -1.9, 95% CI 2-sided [-4.0 to 0.0]
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -0.2, 95% CI 2-sided [-1.4 to 0.8]
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -0.2, 95% CI 2-sided [-1.5 to 1.0]
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-1.2 to 1.5]
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.4, 95% CI 2-sided [-0.4 to 1.4]
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.8 to 1.2]
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -0.4, 95% CI 2-sided [-1.7 to 0.7]
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.4, 95% CI 2-sided [-0.6 to 1.5]
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -0.2, 95% CI 2-sided [-1.3 to 0.7]
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.8 to 1.2]
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 2]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.9, 95% CI 2-sided [-1.2 to 3.0]
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; Serotype 22F; Test type: Superiority — For the 2 serotypes unique to V114, a conclusion of superiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevenar 13™) being >10 percentage points (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen method; Percentage point difference = 94.0, 95% CI 2-sided [91.6 to 95.8]
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; Serotype 33F; Test type: Superiority — [test comment as in outcome 4, analysis 14]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 97.2, 95% CI 2-sided [95.4 to 98.4]

5. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG) 30 Days After Dose 3
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevenar 13™ and 2 serotypes (22F and 33F) unique to V114 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay.
Time Frame: 30 days after Dose 3
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 500 | 525
µg/mL
  Serotype 1 | 1.28 [1.21 to 1.36] | 2.20 [2.08 to 2.34]
  Serotype 3 | 0.85 [0.79 to 0.90] | 0.65 [0.61 to 0.69]
  Serotype 4: number analyzed (Participants) | 500 | 523
  Serotype 4 | 1.41 [1.31 to 1.51] | 2.00 [1.86 to 2.16]
  Serotype 5: number analyzed (Participants) | 500 | 524
  Serotype 5 | 2.08 [1.95 to 2.21] | 3.35 [3.11 to 3.60]
  Serotype 6A: number analyzed (Participants) | 500 | 523
  Serotype 6A | 3.21 [2.97 to 3.47] | 5.36 [4.98 to 5.78]
  Serotype 6B: number analyzed (Participants) | 500 | 523
  Serotype 6B | 4.56 [4.20 to 4.94] | 5.12 [4.71 to 5.57]
  Serotype 7F | 2.78 [2.64 to 2.94] | 3.74 [3.53 to 3.97]
  Serotype 9V: number analyzed (Participants) | 499 | 525
  Serotype 9V | 2.14 [2.02 to 2.27] | 3.07 [2.89 to 3.26]
  Serotype 14: number analyzed (Participants) | 500 | 523
  Serotype 14 | 5.35 [4.93 to 5.80] | 6.83 [6.33 to 7.37]
  Serotype 18C | 2.10 [1.98 to 2.23] | 2.48 [2.33 to 2.65]
  Serotype 19A: number analyzed (Participants) | 500 | 523
  Serotype 19A | 4.74 [4.43 to 5.08] | 6.38 [5.96 to 6.83]
  Serotype 19F: number analyzed (Participants) | 500 | 524
  Serotype 19F | 4.08 [3.82 to 4.36] | 5.18 [4.85 to 5.53]
  Serotype 23F: number analyzed (Participants) | 497 | 521
  Serotype 23F | 1.58 [1.47 to 1.70] | 1.77 [1.64 to 1.91]
  Serotype 22F: number analyzed (Participants) | 500 | 520
  Serotype 22F | 6.06 [5.68 to 6.46] | 0.09 [0.08 to 0.10]
  Serotype 33F: number analyzed (Participants) | 500 | 510
  Serotype 33F | 3.28 [3.06 to 3.51] | 0.07 [0.06 to 0.07]
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Serotype 1; Test type: Non-Inferiority — For the 13 shared serotypes, a conclusion of non-inferiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/Prevenar 13™) being >0.5 (1-sided p-value <0.025); p < 0.001, t-test, 1 sided; GMC ratio = 0.58, 95% CI 2-sided [0.54 to 0.63]
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Serotype 3; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 1.31, 95% CI 2-sided [1.20 to 1.43]
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Serotype 4; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.70, 95% CI 2-sided [0.63 to 0.78]
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Serotype 5; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.62, 95% CI 2-sided [0.56 to 0.68]
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.60, 95% CI 2-sided [0.54 to 0.67]
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.89, 95% CI 2-sided [0.79 to 1.00]
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.74, 95% CI 2-sided [0.69 to 0.81]
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.70, 95% CI 2-sided [0.64 to 0.76]
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Serotype 14; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.78, 95% CI 2-sided [0.70 to 0.87]
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.85, 95% CI 2-sided [0.77 to 0.92]
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.74, 95% CI 2-sided [0.68 to 0.82]
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; Serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.79, 95% CI 2-sided [0.72 to 0.87]
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; Serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p < 0.001, t-test, 1 sided; GMC ratio = 0.90, 95% CI 2-sided [0.81 to 1.00]
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; Serotype 22F; Test type: Superiority — For the 2 serotypes unique to V114, a conclusion of superiority of V114 to Prevenar 13™ is based on the lower bound of the 2- sided 95% CI for the GMC ratio (V114/Prevenar 13™) being >2.0 (1-sided p-value <0.025); p < 0.001, t-test, 1 sided; GMC ratio = 68.34, 95% CI 2-sided [61.73 to 75.65]
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; Serotype 33F; Test type: Superiority — For the 2 serotypes unique to V114, a conclusion of superiority of V114 to Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the GMC ratio (V114/Prevenar 13™) being >2.0 (1-sided p-value <0.025); p < 0.001, t-test, 1 sided; GMC ratio = 48.99, 95% CI 2-sided [44.45 to 54.01]

6. Secondary Outcome: Percentage of Participants Meeting Specified Vaxelis™ Antigen Reponses 30 Days After Dose 3
Description: Antigen-specific response rates in participants administered V114 concomitantly with Vaxelis™ were compared with response rates in participants administered Prevenar 13™ concomitantly with Vaxelis™, and the percentages of participants meeting specified Vaxelis™ antigen responses recorded. Antigens in Vaxelis™ include: diphtheria toxoid, tetanus toxoid, pertussis toxin (PT), pertussis filamentous hemagglutinin (FHA), pertussis fimbriae 2/3 (FIM 2/3), pertussis pertactin (PRN), Haemophilus influenzae type b polyribosylribitol phosphate (Hib-PRP), hepatitis B surface antigen (HBsAg), and poliovirus serotypes 1, 2, and 3.
Time Frame: 30 days after Dose 3
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 514 | 543
Percentage of participants
  Diphtheria toxoid: % ≥0.1 IU/mL | 100.0 | 99.8
  Tetanus toxoid: % ≥0.1 IU/mL | 100.0 | 99.8
  Pertussis - PT: % ≥5 EU/mL | 100.0 | 99.8
  Pertussis - FHA: % ≥5 EU/mL | 100.0 | 99.8
  Pertussis - FIM 2/3: % ≥20 EU/m L | 99.8 | 99.6
  Pertussis - PRN: % ≥5 EU/mL | 99.8 | 99.6
  Hib-PRP: % ≥0.15 μg/mL: number analyzed (Participants) | 495 | 523
  Hib-PRP: % ≥0.15 μg/mL | 96.8 | 97.9
  HBsAg: % ≥10 mIU/mL: number analyzed (Participants) | 495 | 523
  HBsAg: % ≥10 mIU/mL | 99.0 | 99.6
  Poliovirus 1: % w/ Nab ≥1:8 dilution: number analyzed (Participants) | 502 | 529
  Poliovirus 1: % w/ Nab ≥1:8 dilution | 99.8 | 99.8
  Poliovirus 2: % w/ Nab ≥1:8 dilution: number analyzed (Participants) | 499 | 518
  Poliovirus 2: % w/ Nab ≥1:8 dilution | 100.0 | 99.8
  Poliovirus 3: % w/ Nab ≥1:8 dilution: number analyzed (Participants) | 503 | 529
  Poliovirus 3: % w/ Nab ≥1:8 dilution | 100.0 | 100.0
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Diphtheria toxoid; Test type: Non-Inferiority — A conclusion of non-inferiority of Vaxelis™ administered concomitantly with V114 to Vaxelis™ administered concomitantly with Prevenar 13™ is based on the lower bound of the 2-sided 95% CI for the difference in percentages (V114 - Prevenar 13™) being greater than the specified non-inferiority margin (1-sided p-value <0.025); p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Tetanus toxoid; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Pertussis - PT; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Pertussis - FHA; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Pertussis - FIM 2/3; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.8 to 1.2]
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Pertussis - PRN; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.8 to 1.2]
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Hib-PRP; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -1.1, 95% CI 2-sided [-3.3 to 0.9]
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; HBsAg; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -0.6, 95% CI 2-sided [-2.0 to 0.5]
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Poliovirus 1; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = -0.0, 95% CI 2-sided [-0.9 to 0.9]
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Poliovirus 2; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.2, 95% CI 2-sided [-0.6 to 1.1]
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Poliovirus 3; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p < 0.001, Miettinen & Nurminen method; Percentage point difference = 0.0, 95% CI 2-sided [-0.8 to 0.7]

7. Secondary Outcome: Percentage of Participants Meeting Serotype-specific IgG Threshold Value of ≥0.35 μg/mL 30 Days After Dose 2
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevenar 13™ and 2 serotypes (22F and 33F) unique to V114 were quantitated from participants' sera by a multiplex ECL assay. Immunoglobulin G for the 15 serotypes contained in V114 vaccine was determined using a PnECL assay.
Time Frame: 30 days after Dose 2
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 505 | 499
Percentage of participants
  Serotype 1 | 97.2 | 98.2
  Serotype 3 | 96.8 | 78.0
  Serotype 4: number analyzed (Participants) | 505 | 498
  Serotype 4 | 97.6 | 98.2
  Serotype 5: number analyzed (Participants) | 505 | 498
  Serotype 5 | 92.1 | 91.2
  Serotype 6A: number analyzed (Participants) | 505 | 498
  Serotype 6A | 77.2 | 91.4
  Serotype 6B | 59.0 | 40.3
  Serotype 7F | 98.6 | 99.8
  Serotype 9V: number analyzed (Participants) | 504 | 498
  Serotype 9V | 94.0 | 94.8
  Serotype 14: number analyzed (Participants) | 504 | 498
  Serotype 14 | 96.6 | 96.0
  Serotype 18C | 93.1 | 94.4
  Serotype 19A | 94.1 | 96.6
  Serotype 19F | 98.0 | 99.4
  Serotype 23F: number analyzed (Participants) | 505 | 498
  Serotype 23F | 75.4 | 66.7
  Serotype 22F | 97.8 | 2.0
  Serotype 33F | 49.5 | 1.6

8. Secondary Outcome: GMC of Serotype-specific IgG 30 Days After Dose 2
Description: as for outcome 7
Time Frame: 30 days after Dose 2
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 505 | 499
μg/mL
  Serotype 1 | 1.39 [1.30 to 1.48] | 1.70 [1.60 to 1.81]
  Serotype 3 | 1.10 [1.04 to 1.17] | 0.61 [0.57 to 0.65]
  Serotype 4: number analyzed (Participants) | 505 | 498
  Serotype 4 | 1.74 [1.62 to 1.86] | 1.59 [1.48 to 1.70]
  Serotype 5: number analyzed (Participants) | 505 | 498
  Serotype 5 | 1.14 [1.05 to 1.23] | 1.26 [1.16 to 1.37]
  Serotype 6A: number analyzed (Participants) | 505 | 498
  Serotype 6A | 0.67 [0.61 to 0.73] | 1.53 [1.40 to 1.68]
  Serotype 6B | 0.42 [0.37 to 0.48] | 0.24 [0.22 to 0.27]
  Serotype 7F | 1.69 [1.59 to 1.80] | 2.18 [2.06 to 2.31]
  Serotype 9V: number analyzed (Participants) | 504 | 498
  Serotype 9V | 1.55 [1.43 to 1.68] | 1.55 [1.43 to 1.67]
  Serotype 14: number analyzed (Participants) | 504 | 498
  Serotype 14 | 5.59 [5.09 to 6.13] | 5.48 [4.92 to 6.10]
  Serotype 18C | 1.18 [1.11 to 1.26] | 1.58 [1.46 to 1.70]
  Serotype 19A | 1.70 [1.56 to 1.84] | 2.35 [2.15 to 2.56]
  Serotype 19F | 2.79 [2.59 to 3.01] | 4.04 [3.76 to 4.34]
  Serotype 23F: number analyzed (Participants) | 505 | 498
  Serotype 23F | 0.71 [0.65 to 0.78] | 0.54 [0.49 to 0.59]
  Serotype 22F | 3.16 [2.92 to 3.42] | 0.04 [0.04 to 0.04]
  Serotype 33F | 0.30 [0.27 to 0.34] | 0.04 [0.04 to 0.04]
Statistical Analysis 1: Comparison: V114 vs Prevenar 13™; Serotype 1; Test type: Other; GMC ratio = 0.82, 95% CI 2-sided [0.75 to 0.89]
Statistical Analysis 2: Comparison: V114 vs Prevenar 13™; Serotype 3; Test type: Other; GMC ratio = 1.81, 95% CI 2-sided [1.66 to 1.98]
Statistical Analysis 3: Comparison: V114 vs Prevenar 13™; Serotype 4; Test type: Other; GMC ratio = 1.09, 95% CI 2-sided [0.99 to 1.21]
Statistical Analysis 4: Comparison: V114 vs Prevenar 13™; Serotype 5; Test type: Other; GMC ratio = 0.91, 95% CI 2-sided [0.81 to 1.01]
Statistical Analysis 5: Comparison: V114 vs Prevenar 13™; Serotype 6A; Test type: Other; GMC ratio = 0.44, 95% CI 2-sided [0.38 to 0.50]
Statistical Analysis 6: Comparison: V114 vs Prevenar 13™; Serotype 6B; Test type: Other; GMC ratio = 1.73, 95% CI 2-sided [1.46 to 2.05]
Statistical Analysis 7: Comparison: V114 vs Prevenar 13™; Serotype 7F; Test type: Other; GMC ratio = 0.78, 95% CI 2-sided [0.71 to 0.84]
Statistical Analysis 8: Comparison: V114 vs Prevenar 13™; Serotype 9V; Test type: Other; GMC ratio = 1.00, 95% CI 2-sided [0.90 to 1.12]
Statistical Analysis 9: Comparison: V114 vs Prevenar 13™; Serotype 14; Test type: Other; GMC ratio = 1.02, 95% CI 2-sided [0.89 to 1.18]
Statistical Analysis 10: Comparison: V114 vs Prevenar 13™; Serotype 18C; Test type: Other; GMC ratio = 0.75, 95% CI 2-sided [0.68 to 0.82]
Statistical Analysis 11: Comparison: V114 vs Prevenar 13™; Serotype 19A; Test type: Other; GMC ratio = 0.72, 95% CI 2-sided [0.64 to 0.81]
Statistical Analysis 12: Comparison: V114 vs Prevenar 13™; Serotype 19F; Test type: Other; GMC ratio = 0.69, 95% CI 2-sided [0.62 to 0.77]
Statistical Analysis 13: Comparison: V114 vs Prevenar 13™; Serotype 23F; Test type: Other; GMC ratio = 1.32, 95% CI 2-sided [1.16 to 1.51]
Statistical Analysis 14: Comparison: V114 vs Prevenar 13™; Serotype 22F; Test type: Superiority; GMC ratio = 81.01, 95% CI 2-sided [73.12 to 89.75]
Statistical Analysis 15: Comparison: V114 vs Prevenar 13™; Serotype 33F; Test type: Other; GMC ratio = 7.81, 95% CI 2-sided [6.82 to 8.94]

9. Secondary Outcome: Percentage of Participants Meeting Specified Opsonophagocytic Activity (OPA) Responses 30 Days After Dose 3
Description: OPA for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevenar 13™ and 2 serotypes unique to V114 (22F and 33F) was measured using a multiplex opsonophagocytic assay (MOPA).
Time Frame: 30 days after Dose 3
Population: All randomized participants in the OPA Subset without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and who had sufficient data to perform the analysis for each serotype
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 108 | 95
Percentage of participants
  Serotype 1: % ≥1:9 dilution: number analyzed (Participants) | 108 | 94
  Serotype 1: % ≥1:9 dilution | 98.1 [93.5 to 99.8] | 97.9 [92.5 to 99.7]
  Serotype 3: % ≥1:19 dilution: number analyzed (Participants) | 102 | 92
  Serotype 3: % ≥1:19 dilution | 99.0 [94.7 to 100.0] | 97.8 [92.4 to 99.7]
  Serotype 4: % ≥1:34 dilution: number analyzed (Participants) | 105 | 92
  Serotype 4: % ≥1:34 dilution | 100.0 [96.5 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 5: % ≥1:27 dilution | 100.0 [96.6 to 100.0] | 100.0 [96.2 to 100.0]
  Serotype 6A: % ≥1:232 dilution: number analyzed (Participants) | 100 | 93
  Serotype 6A: % ≥1:232 dilution | 100.0 [96.4 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 6B: % ≥1:40 dilution: number analyzed (Participants) | 106 | 93
  Serotype 6B: % ≥1:40 dilution | 100.0 [96.6 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 7F: % ≥1:61 dilution: number analyzed (Participants) | 106 | 94
  Serotype 7F: % ≥1:61 dilution | 100.0 [96.6 to 100.0] | 100.0 [96.2 to 100.0]
  Serotype 9V: % ≥1:151 dilution: number analyzed (Participants) | 102 | 91
  Serotype 9V: % ≥1:151 dilution | 99.0 [94.7 to 100.0] | 100.0 [96.0 to 100.0]
  Serotype 14: % ≥1:62 dilution: number analyzed (Participants) | 105 | 93
  Serotype 14: % ≥1:62 dilution | 100.0 [96.5 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 18C: % ≥1:115 dilution: number analyzed (Participants) | 104 | 93
  Serotype 18C: % ≥1:115 dilution | 99.0 [94.8 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 19A : % ≥1:31 dilution: number analyzed (Participants) | 108 | 93
  Serotype 19A : % ≥1:31 dilution | 100.0 [96.6 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 19F: % ≥1:113 dilution: number analyzed (Participants) | 104 | 92
  Serotype 19F: % ≥1:113 dilution | 100.0 [96.5 to 100.0] | 100.0 [96.1 to 100.0]
  Serotype 23F: % ≥1:55 dilution: number analyzed (Participants) | 104 | 91
  Serotype 23F: % ≥1:55 dilution | 100.0 [96.5 to 100.0] | 100.0 [96.0 to 100.0]
  Serotype 22F: % ≥1:15 dilution: number analyzed (Participants) | 104 | 91
  Serotype 22F: % ≥1:15 dilution | 100.0 [96.5 to 100.0] | 26.4 [17.7 to 36.7]
  Serotype 33F: % ≥1:20 dilution: number analyzed (Participants) | 105 | 95
  Serotype 33F: % ≥1:20 dilution | 100.0 [96.5 to 100.0] | 98.9 [94.3 to 100.0]

10. Secondary Outcome: Geometric Mean Titers (GMTs) of Serotype-specific OPA 30 Days After Dose 3
Description: Sera from participants was used to measure GMT of the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevenar 13™ and 2 serotypes unique to V114 (22F and 33F) was determined using a MOPA.
Time Frame: 30 days after Dose 3
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | V114 | Prevenar 13™
Number analyzed (Participants) | 108 | 95
Titer
  Serotype 1: number analyzed (Participants) | 108 | 94
  Serotype 1 | 152.2 [122.6 to 189.0] | 184.0 [147.2 to 230.0]
  Serotype 3: number analyzed (Participants) | 102 | 92
  Serotype 3 | 320.4 [266.9 to 384.8] | 296.2 [245.5 to 357.3]
  Serotype 4: number analyzed (Participants) | 105 | 92
  Serotype 4 | 2290.8 [1856.9 to 2826.1] | 2842.0 [2404.6 to 3359.0]
  Serotype 5 | 855.5 [699.9 to 1045.7] | 1024.5 [850.5 to 1234.0]
  Serotype 6A: number analyzed (Participants) | 100 | 93
  Serotype 6A | 3316.8 [2828.4 to 3889.5] | 4649.1 [3951.6 to 5469.7]
  Serotype 6B: number analyzed (Participants) | 106 | 93
  Serotype 6B | 2691.6 [2244.4 to 3227.8] | 2658.7 [2234.2 to 3163.8]
  Serotype 7F: number analyzed (Participants) | 106 | 94
  Serotype 7F | 5819.2 [4985.3 to 6792.7] | 7839.0 [6786.9 to 9054.2]
  Serotype 9V: number analyzed (Participants) | 102 | 91
  Serotype 9V | 2192.1 [1807.8 to 2658.1] | 2745.1 [2284.2 to 3298.9]
  Serotype 14: number analyzed (Participants) | 105 | 93
  Serotype 14 | 3449.4 [2803.1 to 4244.7] | 2360.2 [1972.4 to 2824.3]
  Serotype 18C: number analyzed (Participants) | 104 | 93
  Serotype 18C | 2203.1 [1872.6 to 2592.1] | 2003.4 [1725.7 to 2325.7]
  Serotype 19A: number analyzed (Participants) | 108 | 93
  Serotype 19A | 2839.1 [2455.2 to 3282.9] | 3843.6 [3366.9 to 4387.8]
  Serotype 19F: number analyzed (Participants) | 104 | 92
  Serotype 19F | 1748.4 [1469.8 to 2079.7] | 2067.0 [1800.1 to 2373.4]
  Serotype 23F: number analyzed (Participants) | 104 | 91
  Serotype 23F | 3650.2 [3041.3 to 4381.0] | 6776.2 [5344.0 to 8592.3]
  Serotype 22F: number analyzed (Participants) | 104 | 91
  Serotype 22F | 2927.9 [2547.0 to 3365.7] | 29.3 [17.8 to 48.4]
  Serotype 33F: number analyzed (Participants) | 105 | 95
  Serotype 33F | 13334.7 [11334.6 to 15687.7] | 1557.9 [1227.3 to 1977.5]

ADVERSE EVENTS:
Time Frame: Non-serious AEs: up to 14 days after each vaccination dose; serious AEs and deaths (all causes): up to approximately 6 months after Dose 3 (up to approximately 16 months)
Description: The safety analysis population included all randomized participants who received at least 1 dose of study vaccination. The analysis population for All-Cause Mortality included all randomized participants.
Arm/Group | V114 | Prevenar 13™
All-Cause Mortality (participants affected / at risk) | 1/595 | 0/596
Serious Adverse Events (participants affected / at risk) | 30/595 | 28/594
Other Adverse Events (participants affected / at risk) | 590/595 | 592/594
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=595) | Prevenar 13™ (N=594)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 3 (3)
Pertussis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (5)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Infantile spasms (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=595) | Prevenar 13™ (N=594)
Diarrhoea (Gastrointestinal disorders) | 69 (82) | 70 (89)
Teething (Gastrointestinal disorders) | 47 (60) | 50 (67)
Vomiting (Gastrointestinal disorders) | 31 (38) | 38 (41)
Injection site erythema (General disorders) | 357 (613) | 389 (658)
Injection site induration (General disorders) | 339 (658) | 351 (679)
Injection site pain (General disorders) | 375 (646) | 354 (595)
Injection site swelling (General disorders) | 276 (444) | 262 (417)
Pyrexia (General disorders) | 318 (728) | 330 (762)
Nasopharyngitis (Infections and infestations) | 70 (80) | 84 (101)
Body temperature increased (Investigations) | 51 (74) | 61 (91)
Decreased appetite (Metabolism and nutrition disorders) | 326 (632) | 346 (686)
Somnolence (Nervous system disorders) | 460 (1118) | 463 (1085)
Irritability (Psychiatric disorders) | 573 (2266) | 559 (2304)
Urticaria (Skin and subcutaneous tissue disorders) | 100 (130) | 127 (173)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT04016714/Prot_SAP_000.pdf